CLINICAL TRIAL: NCT00695357
Title: Opinion of Patients Under Treatment That Meets the Criteria of New Treatment Strategy According to GINA 2006
Acronym: EPAGGELIA
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Pontikis Panagiotis, MD, Medical and Regulatory Director, AstraZeneca Greece, AstraZeneca SA, Greece
Other Study IDs: NIS-RGR-DUM-2008/1
Record Dates: First submitted 2008-06-09; First posted 2008-06-11 (Estimated); Last update posted 2009-04-30 (Estimated); Status verified 2009-04

CONDITIONS: New Strategies; GINA 2006; Patient Opinion
Keywords: Asthma treatment; GINA 2006; patient perception

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Cross-sectional, one visit study. All the data will be collected through questionnaires. Descriptives statistics will be applied to the data. 832 patients will participate to the study and 104 physicians.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with persistent asthma (GINA 2005) for at least 6 months before entering the study
* Patients who are under treatment according to the new strategies described in GINA 2006 for at least 3 months before entering the study

Exclusion Criteria:

* Patients who are not willing to sign the Informed Consent Form
* COPD Patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care
Sampling Method: Non-Probability Sample
Enrollment: 832 (Estimated)
Dates: Start 2008-04; Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Percentage (%) of Asthma treatment satisfaction and control grading | single visit / once

SECONDARY OUTCOMES:
Rate of treatment compliance | single visit / once
Patients quality of life under treatment | single visit / once

CONTACTS AND LOCATIONS:
Overall Officials: Zachariadis Manolis, MD, Principal Investigator — Euroclinic, Athens, Greece
Locations (31):
- Greece (31):
  - Research Site, Aleksandroupoli
  - Research Site, Amaliáda
  - Research Site, Argos
  - Research Site, Arta
  - Research Site, Athens
  - Research Site, Chania
  - Research Site, Drama
  - Research Site, Githio
  - Research Site, Goúnari
  - Research Site, Heraklion
  - Research Site, Imathia
  - Research Site, Ioannina
  - Research Site, Kalamata
  - Research Site, Katerini
  - Research Site, Kavala
  - Research Site, Komotini
  - Research Site, Lamia
  - Research Site, Larissa
  - Research Site, Nafpaktos
  - Research Site, Neapoli
  - Research Site, Pátrai
  - Research Site, Pírgos
  - Research Site, Rafina
  - Research Site, Serres
  - Research Site, Sparti
  - Research Site, Thessaloniki
  - Research Site, Trikala
  - Research Site, Tripoli
  - Research Site, Véria
  - Research Site, Volos
  - Research Site, Xalkida